CLINICAL TRIAL: NCT04016155
Title: Randomised Controlled Trial of Flash Glucose Monitoring in Reduction of Hypoglycaemia in Diabetes Patients with Chronic Kidney Disease
Brief Title: Flash Glucose Monitoring in Reduction of Hypoglycaemia in Diabetic Patients with Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Elaine Chow, Clinical Lecturer, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FlashDKD
Record Dates: First submitted 2019-06-25; First posted 2019-07-11 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2021-01

CONDITIONS: Diabetes with Diabetic Chronic Kidney Disease (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMBG (Active Comparator): Patients use their own glucometers as control
  Interventions: Device: Patient Own SMBG
- Flash CGMS (Experimental)
  Interventions: Device: Abbott FreeStyle Libre

INTERVENTIONS:
Device: Abbott FreeStyle Libre — Flash CGMS
  Arms: Flash CGMS
Device: Patient Own SMBG — Market SMBG
  Arms: SMBG

SUMMARY:
This will be a single centre study at the Prince of Wales Hospital, Hong Kong. Patients will be identified from an existing registry of diabetes patients with CKD. Potential subjects will be identified from patients attending diabetes, general medical and renal clinics.

Following informed consent, patients will undergo screening where baseline HbA1c, renal function will be measured along withcomprehensive medical and drug history to confirm eligibility. All eligible patients will be fitted with a blinded CGM (Medtronic iPro2 professional CGM) on week-1 for baseline glucose profiles for capturing baseline CGM profile. In case of blinded CGM sensor loss or malfunction, the sensor will be replaced once. Patients with at least 50% sensor data during the blinded wear period will proceed to randomization.

At week 0, patients will be randomized to the flash glucose monitoring or SMBG. Both groups will receive standardised education on diabetes self-management, prevention and treatment of hypoglycaemia. This will be accordance with the usual practice at the study site. In the FGM group, patients will receive training on insertion, operation of the device with access to the device software for viewing of ambulatory glucose profiles. Patients will be advised to confirm blood glucose readings with SMBG in the event of hypoglycaemic symptoms, if FGM displays glucose <3.9mmol or in event of glucose instability.

Patients randomized to the control group will perform SMBG using dedicated blood glucose meter at least twice daily.

Blinded CGM will again be worn in both groups at week 16 for assessment of primary and secondary outcomes.

Subjects will compete a hypoglycaemia diary for documenting symptomatic or asymptomatic hypoglycaemia during the study period.

Questionnaires on hypoglycaemia unawarenesss, fear of hypoglycaemia and patient-reported outcomes will be completed at baseline, week 8 and week 16 in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Type I or II diabetes mellitus diagnosed for at least 6 months
2. Male or female age ≥ 18 years old and ≤ 75 years old.
3. Women who are not pregnant, lactating or planning a pregnancy during their participation in the clinical study.
4. Patients with CKD stage 3b, 4 or 5 as defined by estimated glomerular filtration rate less than 45ml/min/m2
5. History of at least 1 episode of non-severe or severe hypoglycaemia in the 12 months prior to screening
6. Willingness, ability and commitment to comply with the testing, procedure and follow-up outlined in this protocol including (but not limited to) and use of pre-specified glucose monitoring devices.
7. Willingness to perform SMBG during the study period
8. In the opinion of the investigator, absence of any physical limitations, addictive diseases, or underlying medical conditions (including mental health) that may preclude the patient from being a suitable study candidate.
9. Written informed consent to participate in the study provided by the patient.
10. Willing and capable of use of a flash glucose monitor as judged by the investigator

Exclusion Criteria:

1. HbA1C >8.5% at screening
2. Currently pregnant, as demonstrated by a positive pregnancy test at screening or planning pregnancy. Women of childbearing potential will also be asked to adopt adequate contraceptive measures throughout the study period, and to notify the study staff immediately if discovered pregnant. Participants who are unwilling to comply with these measures will be excluded.
3. Any active acute or chronic disease or condition that, in the opinion of the investigator, might interfere with the performance of this study.
4. Any active acute or chronic infectious disease that, in the opinion of the investigator, would pose an excessive risk to study staff.
5. Current use or recent exposure to any medication that in the opinion of the investigator could have an influence on the patient's ability to participate in this study or on the performance of the test device.
6. Extensive skin changes/diseases that preclude wearing the FGM on normal skin at the proposed application sites (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis).
7. Have a known allergy to medical-grade adhesives
8. Known current or recent alcohol or drug abuse
9. Diabetic ketoacidosis, hyperosmolar hyperglycaemic state or myocardial infarction in the six months prior to screening
10. Patients on renal replacement therapy
11. Currently participating in another investigational study protocol where the testing or results may interfere with study compliance, diagnostic results, or data collection.
12. An identified protected vulnerable patient (including but not limited to those in detention, or a prisoner).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Difference in time in hypoglycaemia | week 16
  Compare the difference in time in hypoglycaemia (<3.9mmol/l) on blinded CGM between intervention and control groups

SECONDARY OUTCOMES:
CGM indices | week 16
  Time-in-range (4-10mmol/l), time-in-hyperglycaemia (>10mmol), low blood glucose index, glycaemic variability (coefficient of variation). These CGM indices are defined in accordance with the latest International Consensus on Use of CGM
Glycated haemoglobin | week 16
  Change in HbA1c
Incidence of hypoglycaemia | week 16
  Numbers of hypoglycaemic episode reported by study subjects
Patient compliance to Flash CGMS | week 16
  Frequency of sensor scans and time duration of sensor wear
Change in Diabetic treatment | week 16
  Physician directed change in diabetes treatment (including insulin dosage)
Patient quality-of-life | week 16
  Measures by questionnaire: Diabetes Distress Scale (DDS; total score from 17-102), comprising 3 subscales namely emotional, physician, regimen / social support. A lower score indicates better outcome.
Hypoglycaemia awareness | 16 weeks
  Measure by questionnaire: Gold Score Hypoglycaemia awareness (Total 7 grading, lowest score indicates better outcome)
Treatment satisfaction | 16 weeks
  Measured by questionnaire: IDTSQs (Total 8 questions with total score 0-48, highest score indicates better outcome)
Fear of hypoglycaemia | 16 weeks
  Measured by questionnaire: Hypoglycemia Fear Survey II (comprising 2 subscales namely behaviour (15 items) and worry (18 items). Each item has 5 categorical selection from "never" to "always".

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Chow, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No